CLINICAL TRIAL: NCT06983210
Title: Multi-center, Open-Label, Single Arm Trial for Evaluation of the Efficacy and Safety in the First Line Combination Therapy of Gemcitabine, Cisplatin and Nivolumab With Additional Pretreatment of AM80 for Urothelial Carcinoma Patients
Brief Title: Clinical Trial of AM80 in Combination With Gemcitabine, Cisplatin, and Nivolumab in Patients With Urothelial Carcinoma
Acronym: GRAPE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nagoya University (Other)
Collaborators: Japan Agency for Medical Research and Development (Other Government); Kyushu University (Other); Chiba University (Other); University of Tsukuba (Other); Kyoto University (Other)
Responsible Party: Principal Investigator, Tomoyasu Sano, Lecturer (Department of Urology), Nagoya University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIKE-1(362003)
Record Dates: First submitted 2025-05-02; First posted 2025-05-21 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Urothelial Carcinoma Bladder; Urothelial Carcinoma of the Renal Pelvis and Ureter; Urothelial Carcinoma Urethra; Urothelial Carcinoma Recurrent
Keywords: urothelial carcinoma; Gemcitabine, Cisplatin and Nivolumab; bladder cancer; renal pelvis cancer; ureteral cancer; urethral cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Ureteral Neoplasms; Urethral Neoplasms | interventions — tamibarotene; Cisplatin

STUDY DESIGN:
Intervention Model Description: In this study, treatment period 1 will consist of one course of 3 weeks (21 days) in principle, and up to 6 courses will be continued. After discontinuation of Treatment Phase 1 (when gemcitabine or cisplatin cannot be continued) or termination of Treatment Phase 1, AM80 and nivolumab will be continued for one course of 4 weeks (28 days) in principle, until either the discontinuation criteria are met or the imaging evaluation at 49 weeks is completed. During the follow-up period, patients will be followed until the last patient completes the imaging evaluation at 49 weeks, with a follow-up survey every 8 weeks until 49 weeks after the first dose of AM80, and a follow-up survey every 12 weeks after 49 weeks after the first dose of AM80, as follow-up survey (1).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MIKE-1 (Experimental): A characteristic pathology of refractory cancers such as advanced urothelial carcinoma is a high proliferation of cancer-associated fibroblasts (CAFs) in the stroma and associated fibrosis. The investigators have previously identified fibroblast-specific meflin as the first functional marker of tumor suppressive CAFs. The investigators hypothesize that increasing the number of mephrin-positive tumor suppressive CAFs may increase the efficacy of ICI. The investigators investigated this in a mouse model of bladder cancer among urothelial carcinomas and confirmed that AM80 administration markedly increased the therapeutic efficacy of ICI. The investigators considered that the efficacy of ICI may be enhanced in patients with urothelial carcinoma when AM80 is administered in combination with ICI.
  Based on the above, The investigators will explore and evaluate the efficacy and confirm the safety of AM80 when administered in combination with nivolumab, gemcitabine, and cisplatin.
  Interventions: Drug: Add-on effect of adding tamivarotene (AM80) to gemcitabine, cisplatin, and nivolumab combination therapy

INTERVENTIONS:
Drug: Add-on effect of adding tamivarotene (AM80) to gemcitabine, cisplatin, and nivolumab combination therapy — To explore the efficacy and safety of the combination of tamivarotene (AM80), gemcitabine, cisplatin, and nivolumab in the treatment of patients with untreated unresectable or recurrent urothelial cancer
  Other Names: AM80

SUMMARY:
【Treatment of Urothelial Carcinoma】 Treatment for urothelial carcinoma includes surgery, chemotherapy (anticancer drugs), and radiation therapy. Chemotherapy is generally used when metastasis has already occurred at diagnosis and surgery is not curative (metastatic urothelial carcinoma) or when the cancer recurs after local therapy such as surgery or radiation therapy (recurrent urothelial carcinoma).

Although there are several recommended treatments for urothelial carcinoma, the options are often limited by side effects and other factors, and these treatments may not be fully effective. Therefore, the development of safer and more effective treatments is desired.

【About the Drugs to be Used in this Clinical Trial】 In this clinical trial, the investigational drug MIKE-1 will be used in combination with nivolumab plus GC (cisplatin gemcitabine), one of the recommended chemotherapy regimens, and subsequently with nivolumab monotherapy for patients with unresectable metastatic or recurrent urothelial cancer. Nivolumab, cisplatin, and gemcitabine are injectable (intravenous infusion), while MIKE-1 is oral.

【Purpose of the Clinical Trial】 The purpose of this clinical trial is to evaluate the efficacy (how much the cancer shrinks or slows down) and safety of the investigational drug MIKE-1 in combination with nivolumab and gemcitabine and cisplatin therapy in patients with untreated unresectable or recurrent urothelial cancer.

DETAILED DESCRIPTION:
【Treatment of urothelial carcinoma】 Treatment for urothelial carcinoma includes surgery, chemotherapy (anticancer agents), and radiation therapy. Chemotherapy is generally used when metastasis has already occurred at the time of diagnosis and surgery is not curative (metastatic urothelial carcinoma), or when cancer has reappeared after local therapy such as surgery or radiation therapy (recurrent urothelial carcinoma).

Pembrolizumab plus enfoltumab vedotin, cisplatin and gemcitabine (GC) plus nivolumab followed by nivolumab alone, or GC followed by avelumab are the recommended standard of care for patients with metastatic or recurrent urothelial carcinoma. The standard of care for recurrent urothelial carcinoma is Although there are several recommended treatments for urothelial carcinoma, the options are often limited by side effects and other factors, and the effectiveness of these treatments may not be sufficient. Therefore, the development of safer and more effective treatments is desired.

Thus, although treatment methods for urothelial carcinoma are gradually advancing, options are often limited by side effects and other factors, and effectiveness is not yet sufficient. Therefore, the development of safer and more effective treatments is desired.

【About the drugs to be used in this clinical trial】 In this clinical trial, the investigational drug "MIKE-1" will be used in combination with "nivolumab + GC (cisplatin and gemcitabine) combination therapy and subsequent nivolumab monotherapy," which is one of the chemotherapy regimens recommended overseas for patients with unresectable metastatic or recurrent urothelial cancer . Nivolumab, cisplatin and gemcitabine are injectable (intravenous infusion) and MIKE-1 is oral.

・ Investigational drug MIKE-1 (AM80) MIKE-1 is a soft capsule formulation containing the active ingredient AM80 (also called tamivarotene), a member of the vitamin A family called synthetic retinoids.

A tablet formulation containing the same active ingredient as MIKE-1 was approved and is currently used in Japan for the treatment of acute promyelocytic leukemia in April 2005 under the trade name Amnolake® Tablets.

Metastatic or recurrent urothelial carcinoma is thought to have many areas surrounding cancer cells called stroma, which makes it difficult for anticancer drugs to reach the cancer cells and thus makes the treatment less effective.

Nagoya University has confirmed in animal studies that AM80 softens cancer stroma, making it easier for anticancer drugs to reach cancer cells. It was also confirmed that when AM80 is used in combination with immune checkpoint inhibitors（ICIs）, immune cells with enhanced functions to attack cancer cells gather in large numbers around the cancer cells, and the tumors become smaller. Based on these results, the investigators planned this clinical trial in the hope that the administration of MIKE-1, whose active ingredient is AM80, in combination with ICIs used for urothelial carcinoma will enhance the effect of tumor reduction.

【Purpose of the Clinical Trial】 The purpose of this study is to evaluate the efficacy (how much the cancer is reduced or slowed down) and safety of the investigational drug MIKE-1 in combination with nivolumab and GC therapy in patients with untreated unresectable or recurrent urothelial carcinoma in the urothelial cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been histologically or cytologically diagnosed with urothelial carcinoma of the renal pelvis, ureter, bladder, or urethra based on the General Rule for Clinical and Pathological Studies on Renal Pelvic, Ureteral and Bladder Cancer, 2nd Edition that cannot be curatively resected or has recurred (diagnosis is not permitted at the site of palliative radiation)
2. Patients who have not received prior treatment for unresectable or recurrent urothelial carcinoma
3. Patients with measurable lesions according to RECIST version 1.1 on the CT at screening
4. Patients with an ECOG PS of 0-1 at screening, who are able to take oral medication
5. Patients who will be expected to survive for 12 weeks or more from the enrollment
6. Patients whose major organ functions at screening meet the following criteria

(1)Neutrophil count: 1,500/uL or more (2)Platelet count: 100,000/uL or more (3)Hb: 9.0 g/dL or more (no red blood cell transfusion within 14 days prior to screening examination) (4)T-Bil: 1.5 times or less than 1.5 times the upper limit of the facility standard value (less than 3.0 mg/dL in the case of Gilbert syndrome) (5)AST and ALT: 3 times or less than 3 times the upper limit of the facility standard value (6)CrCl 50 mL/min or more 7.Patients who have given consent to be treated if any of the following applies:

1. Female patients of childbearing potential who can prevent contraception for 30 days prior to enrollment and for 2 years after the end of AM80 treatment
2. Male patients with partners of childbearing potential, who can use contraception from the start of AM80 administration until 7 months after the end of administration and refrain from donating sperm during the above period 8.Patients aged 18-79 years at the time of consent (regardless of sex) 9.Patients who have received a thorough explanation of this clinical trial and have voluntarily given their written informed consent

Exclusion Criteria:

1. Patients who have previously been treated with drugs such as antibodies targeting PD-1, PD-L1, PD-L2, CTLA-4, OX-40, or CD137
2. Patients who have received any of the following t reatments for urothelial carcinoma:

(1)Perioperative adjuvant therapy for curative resection completed less than 12 months prior to enrollment (2)Intravesical therapy within 28 days prior to enrollment (3)Palliative radiation therapy for measurable lesions within 14 days prior to enrollment 3.Patients who have not recovered from toxicity (Grade 1 or 0 or at baseline) from prior treatment at the time of enrollment; however, enrollment is permitted for those with <= Grade 2 fatigue and alopecia 4.Patients who have participated in other clinical trials within 28 days prior to enrollment (enrollment is permitted if the drug or medical device used in the clinical trial are similar to approved indications, dosage, and administration and do not affect the evalu ation) and who have received their last dose of a drug or other substance used in the current clinical research within the last 28 days 5.Patients with metastasis to the central nervous system or a history or complication of carcinomatous meningitis 6.Patients with multiple cancers whose disease-free interval at the time of registration is less than 3 years (excluding gastrointestinal cancer that was completely resected via endoscopic mucosal resection, completely resected intraepithelial neoplasia of the cervix, localized or presumably cured prostate cancer, completely resected basal/squamous cell carcinoma of the skin, and solid cancers similar to these that have undergone curative treatment and are presumed to be cured) 7.Patients who are taking vitamin A agents or vitam in A-containing supplements at the time of enrollment 8.Patients who have undergone surgery under general anesthesia (excluding diagnostic biopsies) or severe trauma within 28 days prior to enrollment 9.Patients known to have a bleeding tendency or coagulation disorder (e.g., patients with significant in tratumoral bleeding, thromboembolism, or a history or comorbidity of bleeding disorders), and those who require administration of anticoagulants or antiplatelet drugs 10.Patients with active infections requiring systemic administration of antibiotics, antifungals, or antivirals 11.Patients who test positive for hepatitis B surface (HBs) antigen, hepatitis C virus (HCV) antibody and RNA, or HIV antigen or antibody. However, even if the patient is negative to HBs antigen, if the patient is positive to HBs antibody or hepatitis B core (HBc) antibody, the possibility of inclusion should be considered in consultation with a gastroenterologist, if necessary, based on Document 3 of the latest Hepatitis B Treatment Guidelines.

12.Patients with a history of or comorbidity of interstitial lung disease evident on imaging, or those with active non-infectious pneumonitis 13.Patients with autoimmune disease, a history of chronic or recurrent autoimmune disease, or those who have required high-dose systemic corticosteroids (prednisolone equivalent of more than 10 mg/day) or immunosuppressants within 14 days prior to enrollment 14.Patients who require treatment for tuberculosis 15.Patients with clinical symptoms or findings indicating intestinal obstruction requiring intravenous or total parenteral nutrition, and those with risk factors for intestinal perforation (e.g., acute diverticulitis, in traperitoneal abscess, gastrointestinal obstruction, history of abdominal tumor, etc.).

16.Patients with gastrointestinal disorders that may affect the absorption of AM80 17.Patients with a history of severe hypersensitivity or anaphylactic reactions to components of the drugs used in the clinical trial or antibody preparations 18.Patients who received live or attenuated vaccines within 30 days prior to enrollment 19.Patients with serious complications (liver disease , kidney disease, heart disease, lung disease, blood disease, brain disease, etc.) 20.Patients with uncontrolled adrenal insufficiency, Grade 2 or higher hearing impairment, or Grade 2 or higher neuropathy 21.Patients with hypervitaminosis A 22.Lactating female patients (excluding those who agreed to discontinue breastfeeding during the study period and for 6 months after the final dose of A M80) 23.Female patients who are pregnant or have positive pregnancy test results (female patients who have had a period within 12 months prior to enrollment and may be pregnant will be subjected to a pregnancy test. Female patients who have not had a period within 12 months but whose pregnancy cannot be ruled out due to reasons such as chemical menopause will also be subjected to a pregnancy test) 24.Patients who are otherwise deemed inappropriate for participation in this clinical trial by the principal investigator or sub-investigator

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Response rate (RR) | Time from the start of treatment (day 1) to the confirmation of complete response (CR: complete disappearance of tumor) or partial response (PR: reduction of tumor by a certain percentage or more). (Average 18 weeks)
  Response rate (RR): determined by the investigator or sub-investigator at the site.
  Tumor shrinkage by the best overall response based on the RECIST criteria will be determined by CT scan at each time point. For the same subject, the same imaging method used to evaluate measurable lesions at screening (e.g., the same contrast method) will be used during the study period in principle. The evaluation on each visit day should be performed by the same evaluator as much as possible to ensure internal consistency between each visit day. The response rate is calculated as the ratio of the total number of subjects with complete response (CR) and partial response (PR). CR or PR shall require "confirmation of efficacy".

SECONDARY OUTCOMES:
Overall survival | Time from day 1 of AM80 administration to death. (Average 49 weeks)
  Overall survival is defined as the period beginning on the date of AM80 administration and ending on the date of death from any cause.
  For cases that are alive at the cutoff point, the last date of confirmed survival is used as the cutoff date. In the case of untraceable cases, the cutoff date is the last date of confirmed survival before the cutoff.
Progression free survival | Time from day 1 of AM80 administration to the date of confirmed progression. (Average 49 weeks)
  Progression" in the evaluation of progression-free survival is defined as Progressive Disease (PD) in the overall efficacy. Progression-free survival is defined as the time to the cut-off point for survivors who have not experienced progression by the time the last patient completes the imaging evaluation at 49 weeks post-treatment (cut-off point). Unfollow-up will be terminated on the date of the last confirmation that there was no progression. For subjects who have started post-treatment without progression, the cut-off date is the date of the last confirmation that there was no progression before the start of post-treatment. However, if nivolumab is continued after completion of study treatment, it will be treated as post-treatment, but will not be censored in the calculation of progression-free survival. If post-treatment other than nivolumab is subsequently started, it will be censored on the last date of confirmation that no progression occurred before that date.
Duration of Response | Time since initiation of treatment from the time PR or CR was first identified to the date of tumor recurrence. (Average 49 weeks)
  The duration of response is the period from the start of AM80 administration to the first date of objective confirmation of tumor recurrence or progression of disease from the time of first confirmation of CR or PR in the evaluation of overall efficacy from the start of AM80 administration in cases in which the best overall response was evaluated as CR or PR. The duration of complete response is the period from the start of AM80 administration and the first confirmed CR in the assessment of overall response to the first objectively confirmed date of tumor recurrence. Duration of response and duration of complete response will be evaluated based on the determination by RECIST evaluation, respectively.
  If no progression of disease is observed at the cut-off time point, the study is terminated on the last date when disease progression is confirmed. For subjects who have started post-treatment without progression, the cut-off date will be the last date of confirmation that there was no p

CONTACTS AND LOCATIONS:
Overall Officials: Syusuke Akamatsu, Principal Investigator — Nagoya University Hospital
Locations (1):
- Nagoya University Hospital, Nagoya, Aichi-ken, Japan

IPD SHARING:
Plan to Share IPD: Yes
The secondary use of all IPD datas that underlie results in a publication excluding personal information will be acceptable after publication of results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 3 years after the publication of results.
Access Criteria: If the principal investigator, clinical trial office, main stakeholder conclude that secondary use of individual data obtained in this clinical trial is beneficial for additional analysis, the secondary use of data excluding personal information will be acceptable after publication of results.

REFERENCES:
- [Background] Owaki T, Iida T, Miyai Y, Kato K, Hase T, Ishii M, Ando R, Hinohara K, Akashi T, Mizutani Y, Ishikawa T, Mii S, Shiraki Y, Esaki N, Yamamoto M, Tsukamoto T, Nomura S, Murakami T, Takahashi M, Yuguchi Y, Maeda M, Sano T, Sassa N, Matsukawa Y, Kawashima H, Akamatsu S, Enomoto A. Synthetic retinoid-mediated preconditioning of cancer-associated fibroblasts and macrophages improves cancer response to immune checkpoint blockade. Br J Cancer. 2024 Jul;131(2):372-386. doi: 10.1038/s41416-024-02734-3. Epub 2024 Jun 7. PMID 38849479